CLINICAL TRIAL: NCT04480151
Title: ExtraCorporeal Life Support (ECLS) Versus IMPELLA™ Pump as Bridge to Left Ventricular Assist Device
Brief Title: ECLS Versus IMPELLA™ as Bridge to LVAD (ECI-BLAD)
Acronym: ECI-BLAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/37
Record Dates: First submitted 2020-07-13; First posted 2020-07-21 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Cardiogenic Shock; End-stage Heart Failure
Keywords: cardiogenic shock; end stage heart failure; bridge to bridge; bridge to decision; left ventricular assist device; IMPELLA™; ECLS
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMPELLA™ alone as bridge to LVAD: patients assisted by IMPELLA™ pump alone during the days preceding the implantation of long term LVAD (at least 48 hours for patients for whom an ECLS was previously used)
  Interventions: Other: standard of care
- ECLS alone or with IMPELLA™ as bridge to LVAD: patients assisted by ECLS (ExtraCorporeal life support) alone or simultaneously with IMPELLA™ until the implantation of LVAD
  Interventions: Other: standard of care

INTERVENTIONS:
Other: standard of care — retrospective study: standard of care

SUMMARY:
In this retrospective observational multicenter study the authors tested the hypothesis that the use of IMPELLA™ pump as bridge to bridge, by giving the opportunity of active rehabilitation, should improve patient's outcomes after the implantation of Left Ventricular Assist Device (LVAD).

DETAILED DESCRIPTION:
End stage heart failure patients admitted in Intensive Care Unit (ICU) for refractory cardiogenic shock requiring short-term mechanical circulatory support as a bridge to a long-term LVAD might benefit from early mobilization and rehabilitation with IMPELLA™ inserted via the axillary artery. The aim of this study is to compare the early rehabilitation and outcomes after LVAD implantation between patients previously treated by IMPELLA™ or ExtraCorporeal Life Support (ECLS)

ELIGIBILITY:
Inclusion Criteria:

* patients supported with IMPELLA™ or ECLS for refractory cardiogenic shock as a bridge to long duration LVAD

Exclusion Criteria:

* Patient refusing to give access to their medical chart
* Guardianship and curactorship
* Deprived of liberty
* short term mechanical circulatory system weaned before LVAD implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients implanted by IMPELLA™ pump or ECLS as a bridge to long duration LVAD between January 2012 and December 2018 in five university hospital centers.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
Proportion of patients alive in the surgery ward, not requiring intravenous access and walking (John Hopkins highest level of mobility (JH-HLM) scale = 8 at 30 days after the LVAD implantation | Day 30 after Left Ventricular Assist Device (LVAD) implantation
  Proportion of patients alive in the surgery ward, not requiring intravenous access and walking (John Hopkins highest level of mobility (JH-HLM) scale = 8) at 30 days after the LVAD implantation

SECONDARY OUTCOMES:
Complication and rehabilitation under Short-term Mechanical Circulatory support | The day of Left Ventricular Assist Device (LVAD) implantation
  Duration of support, bleeding, hemolysis, surgical re-exploration, thombus, renal replacement therapy, blood products transfusion, stroke, tracheal extubation, mobilization (chair, walking and ergometry)
Organ dysfunction before LVAD implantation | The day before LVAD implantation
  Need for mechanical ventilation, Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
complication Under LVAD | The day of Intensive Care Unit (ICU) discharge
  bleeding, right ventricular dysfunction, vasoplegia
SOFA score | The day of Short Term Mechanical Circulatory Support (STMCS) implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
SOFA score | The day of LVAD implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
SOFA score | Day 1 post LVAD implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
SOFA score | Day 3 post LVAD implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
SOFA score | Day 5 post LVAD implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
SOFA score | Day 7 post LVAD implantation
  Organ dysfunction assessed by Sequential Organ Failure Assessment (SOFA) score [0= best outcome to 24 = worst outcome]
Vital status | 1 month after LVAD implantation
  mortality after LVAD implantation
Vital status | 3 months after LVAD implantation
  mortality after LVAD implantation
Vital status | 6 months after LVAD implantation
  mortality after LVAD implantation
length of stay | up to Intensive Care Unit (ICU) discharge (not more than 6 months after LVAD implantation)
  Intensive Care Unit length of stay
length of stay | up to hospital discharge (not more than 6 months after LVAD implantation)
  hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre OUATTARA, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (5):
- France (5):
  - CHU de Dijon-Bourgoigne, Dijon
  - CHU de Montpellier, Montpellier
  - CHU de Bordeaux, Pessac
  - CHU de Rennes, Rennes
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No